CLINICAL TRIAL: NCT05640388
Title: An Exploratory, Comparative and Multicentric Study, to Evaluate the Effect of the RV3278A - ET0943 on the Host/Micro-organism Relationships in Acneic Subjects
Brief Title: Assessment of a Cosmetic Product Effect on the Host/Microorganism Relationship in Acneic Subjects
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV3278A20200403
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Acne
Keywords: Comedones; Lipids; Blackheads; Host/Microorganism Relationship; Micro comedones
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Sebum and comedones constituents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RV3278A arm : Treated group: This group will receive the RV3278A - ET0943 product
  Interventions: Other: RV3278A - ET0943 cosmetic product
- RV4632A arm : Control group: This group will receive the RV4632A - RY1845 product
  Interventions: Other: RV4632A - RY1845 cosmetic product

INTERVENTIONS:
Other: RV3278A - ET0943 cosmetic product — RV3278A - ET0943 study product is applied twice a day on the face during the whole study.
  Groups: RV3278A arm : Treated group
Other: RV4632A - RY1845 cosmetic product — RV4632A - RY1845 study product must be applied only in case of sensation of skin discomfort
  Groups: RV4632A arm : Control group

SUMMARY:
The aim of the study is to understand the structural and functional modifications of the host, the microorganisms, and their interactions (host/microorganism relationship) before and after the RV3278A - ET0943 product application

ELIGIBILITY:
Inclusion Criteria:

1. Related to the population:

   - Subject aged between 12 to 25 years included
2. Related to diseases:

   * Subject having acne lesions on the face, with GEA (Global Acne Evaluation) score on the face is assessed as 2 (mild) or as 3 (moderate), on a scale ranged from 0 (clear- no lesion) to 5 (very severe)
   * Subject having at least 20 open-comedones of about 1 mm in diameter on the face and possibly extractable
   * Subject having a predominance of non-inflammatory acne lesions

Exclusion Criteria:

1. Related to diseases:

   * Subject having comedones only on the nose wings
   * Subject with any other dermatological disease than acne or skin characteristics (like scar, tatoo) on the face liable to interfere with the study according to the investigator's assessment
   * Subject with an acute or chronic disease, or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
   * Severe form of acne (Acne conglobata, Acne fulminans or nodulokystic acne) or acneiform induced rashes according to the investigator's assessment
   * Clinical signs of a hormonal dysfunction or of a hyperandrogenism
   * Solar erythema on the face due to excessive UV exposur
2. Related to the treatments/products:

   * Any previous/concomitant treatment or product considered by the Investigator liable to interfere with the study data or incompatible with the study requirements or hazardous for the subject

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects are enrolled during their usual medical care and/or from the database of the investigational sites.
  The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the study.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Effect of the RV3278A on acne severity | Change from baseline to 2 months
  Global Evaluation Acne (GEA), on a 6-point scale 0: Clear. No lesions
  1. Almost clear, Almost no lesions
  2. Mild
  3. Moderate
  4. Severe
  5. Very severe
Effect of the RV3278A on inflammatory and retentionnal lesions | Change from baseline to 2 months
  Quantification of inflammatory and retentionnal lesions from image analysis
Effect of the RV3278A on microorganisms | Change from baseline to 2 months, for each group
  Quantitative analysis by ddPCR (droplet digital Polymerase Chain Reaction) from comedones samples
Effect of the RV3278A on microorganisms | Change from baseline to 2 months
  Qualitative analysis by 2 and 3-dimensional electron microscopy from comedones samples
Effect of the RV3278A on metabolites | Change from baseline to 1 month
  Metagenomic analysis on comedones samples
Effect of the RV3278A on lipids | Change from baseline to 2 months
  Lipids PCR (Polymerase Chain Reaction) analysis done by SpiderMass tool from cigarette paper and comedones samples
Effect of the RV3278A on lipids | Change from baseline to 2 months
  Qualitative analysis by 2 and 3-dimensional electron microscopy from comedones samples
Effect of the RV3278A on hyperkeratosis | Change from baseline to 2 months
  Qualitative analysis by 2 and 3-dimensional electron microscopy from comedones samples
RV3278A product tolerance | From Day 1 to 2 months
  Adverse events occurrence will be determined by the subject's / parent(s) or guardian(s) spontaneous reporting, the investigator's non-leading questioning, and his/her clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pascal REYGAGNE, Principal Investigator — Centre de Santé Sabouraud
Locations (2):
- France (2):
  - Centre de santé SABOURAUD C.E.P.C, Paris
  - Centre de Recherche sur la Peau, Toulouse